CLINICAL TRIAL: NCT02493686
Title: Age Dependence of Audiometric Bone Conduction Threshold in Normal Hearing Subjects
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PR_16_09_2014
Record Dates: First submitted 2015-06-02; First posted 2015-07-09 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2015-11

CONDITIONS: Air Bone Gap
MeSH Terms: interventions — Audiometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: audiogram — hearing test

SUMMARY:
Examination of the bone conduction of persons which according to the pure tone audiogram have a normal age related hearing threshold in the air conduction.

ELIGIBILITY:
Inclusion Criteria:

* All pure tone audiograms recorded and available in the system from the beginning of measurement as follows:
* age related normal hearing threshold level with air conducted pure tone audiogram

Exclusion Criteria:

* age younger than 20 years
* if inclusion criteria not given

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons which have a normal hearing threshold level in the airconduction.
Sampling Method: Non-Probability Sample
Enrollment: 1093 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Bone conduction Threshold/ Air bone gap in normal hearing subject in relation to age | 1960 - 2014 (54 years)
  from the initial establishment of the database until collection of the data

SECONDARY OUTCOMES:
Air bone gap changes in individuals who have received more than one Audiogram | 1960 - 2014 (54 years)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Probst, Prof., Study Director — University Hospital Zurich, clinic othorhinolaryngology, 8091 Zurich